CLINICAL TRIAL: NCT07295405
Title: Effect of Water Temperature on Bowel Cleansing Quality: A Prospective Observational Study
Brief Title: Water Temperature and Bowel Cleansing Quality
Status: Completed | Type: Observational
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Nurettin Şahin, Consultant General Surgeon, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Other Study IDs: Bakırkoy Sadi konuk trials
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Colonoscopy (Procedure)
Keywords: Colonoscopy; Bowel Preparation; Water Temperature; Boston Bowel Preparation Scale

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Observational study The aim of this observational study is to investigate the effect of water temperature used during pre-colonoscopy bowel preparation on the quality of bowel cleansing. The primary research question to be addressed is as follows: Which water temperature results in better bowel cleansing quality? For this purpose, patients will be divided into two groups based on the use of warm water or cold water, and the quality of bowel preparation will be compared between the groups.

DETAILED DESCRIPTION:
The aim of this observational study is to investigate the effect of water temperature used during pre-colonoscopy bowel preparation on the quality of bowel cleansing. The primary research question to be addressed is as follows: Which water temperature results in better bowel cleansing quality? For this purpose, patients will be divided into two groups based on the use of warm water or cold water, and the quality of bowel preparation will be compared between the groups.

ELIGIBILITY:
Inclusion Criteria: -Patients aged ≥ 18 years undergoing elective colonoscopy -Ability to provide informed consent -Planned bowel preparation using water-based regimens -No contraindication to warm or cold water intake

Exclusion Criteria: - Emergency colonoscopy -History of inflammatory bowel disease -Prior colorectal surgery -Severe heart failure, renal failure, or electrolyte imbalance -Pregnancy -Inability to complete bowel preparation protocol -Use of additional laxatives outside the study protocol

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted to the general surgery endoscopy clinic of a tertiary-care hospital for colonoscopy
Sampling Method: Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
quality of bowel preparation | 01.02.2025-01.07.2025
  The quality of bowel preparation will be assessed using the Boston Bowel Preparation Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Nurettin Şahin, MD, Principal Investigator — Bakırköy Dr. Sadi Konuk Training and Research Hospital
Locations (1):
- Bakırköy Dr. Sadi Konuk Training and Research Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
All study data will be retained by the principal investigator and may be shared when required.

REFERENCES:
- [Result] Shahini E, Sinagra E, Vitello A, Ranaldo R, Contaldo A, Facciorusso A, Maida M. Factors affecting the quality of bowel preparation for colonoscopy in hard-to-prepare patients: Evidence from the literature. World J Gastroenterol. 2023 Mar 21;29(11):1685-1707. doi: 10.3748/wjg.v29.i11.1685. PMID 37077514